CLINICAL TRIAL: NCT06125171
Title: A Phase II Clinical Trial of Tucidinostat in Combination With Apatinib in Patients With Relapsed or Refractory Osteosarcoma
Brief Title: Tucidinostat Plus Apatinib for Advanced Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q54
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat+Apatinib (Experimental)
  Interventions: Drug: Tucidinostat, Apatinib

INTERVENTIONS:
Drug: Tucidinostat, Apatinib — Tucidinostat:
  age≥18years, 30mg, po., biw, q4w; age≥10years，<18years，0.5mg/kg, biw, q4w
  Apatinib:
  BSA≥1.2m^2, 500mg, qd, q4w BSA<1.2m^2, 250mg, qd, q4w

SUMMARY:
This phase II study was designed to assess the efficacy and safety of the combination of Apatinib, Tucidinostat (chidamide), a histone deacetylase inhibitor in relapsed or refractory osteosarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥10 years, ≤ 75 years;
2. Histologically confirmed Advanced classic osteosarcoma with unresectable recurrence or metastatic disease ；
3. Prior treatment consisted of standard chemotherapy agents including doxorubicin, cisplatin, methotrexate, and ifosfamide;
4. Eastern Collaborative Oncology Group (ECOG) 0~2；
5. Tumor size is measurable according to RECIST1.1 criteria；
6. Adequate organ function；
7. Life expectancy is more than 3 months；
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Previously exposed to histone deacetylase inhibitors or angiogenesis inhibitors;
2. Urine protein≥ ++;
3. FBG>10mmol/L;
4. Uncontrolled blodd pressure (ystolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg);
5. Known active CNS metastases and/or carcinomatous meningitis;
6. Not able to take medicine orally;
7. Coagulant function abnormality (PT>16s, APTT> 43s, TT>21s, FIB）<2g/L);
8. Uncontrolled clinically significant systemic diseases, including active infection, unstable angina, angina occurred within 3 months,≥ NYHA II congestive heart failure, myocardial infarction occurred within 6 months, severe arrhythmia, liver, kidney, or metabolic disease;
9. Major surgery received or severe traumatic injury, fracture, or ulcer occurred within 4 weeks of the first dose of study medication.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival rate | 6 months
  The proportion of patients who did not experience disease progression or die from disease progression within 6 months from the treatment

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Time from treatment until disease progression or death
Objective Response Rate（ORR） | 2 years
  Objective Response Rate（ORR）by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）
Disease Control Rate （DCR） | 2 years
  the total proportion of patients with complete response（CR）, partial response（PR）and stable disease（SD）
Overall survival(OS) | 2 years
  Time from treatment until death from any cause

IPD SHARING:
Plan to Share IPD: No